CLINICAL TRIAL: NCT01357187
Title: An Evaluation of the Effect of the AmnioFix™ Amniotic Membrane Allograft on Scar Tissue and Adhesions in Patients Undergoing Posterior Instrumentation Removal
Brief Title: An Evaluation of the Effect of the AmnioFix Amniotic Membrane Allograft in Patients Undergoing Posterior Instrumentation Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFPIR001
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2014-06

CONDITIONS: Adhesions of Soft Tissue
Keywords: Lumbar pathology; requiring elective lumbar interbody fusion

ARMS (2):
- Control (Other)
  Interventions: Other: Scheduled removal of posterior instrumentation without AmnioFix
- Treatment (Experimental)
  Interventions: Other: Scheduled removal of posterior instrumentation with AmnioFix

INTERVENTIONS:
Other: Scheduled removal of posterior instrumentation with AmnioFix
  Arms: Treatment
Other: Scheduled removal of posterior instrumentation without AmnioFix
  Arms: Control

SUMMARY:
The objective of this study is to evaluate the clinical effectiveness of AmnioFix™ in the reduction of the tenacity and frequency of soft tissue adhesions during the removal of segmental posterior lumbar instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Diagnosed with lumbar pathology requiring elective lumbar interbody fusion
* Willingness to comply to follow-up examinations and diagnostic imaging procedures
* Ability to give full written informed consent

Exclusion Criteria:

* Previous surgical procedure performed at same site
* Sign or symptoms of other disease which could result in allograft failure
* Require a corpectomy
* Participating in another drug or device clinical trial
* Pregnant or may become pregnant during the study
* Prisoner
* Involved in workmen's compensation or other litigation relative to a spine injury
* Past medical history of allograft implantation which resulted in graft failure
* Any condition requiring treatment above the normal standard of care
* Currently taking medications which could affect graft incorporation (supervising physicians discretion)
* Auto-Immune disease
* Renal failure
* Failure to sign or understand informed consent information
* History of drug and/or alcohol abuse
* Allergic to aminoglycosides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Tenacity and frequency of soft tissue adhesion | At the time of removal of segmental posterior lumbar instrumentation

SECONDARY OUTCOMES:
Presence and extent of scar tissue using histological analysis of the lumbar tissue adjacent to the surgical site | At the time of removal of segmental posterior lumbar instrumentation
Number of intra-operative complications | At the time of removal of segmental posterior lumbar instrumentation

CONTACTS AND LOCATIONS:
Overall Officials: Brian Subach, MD, Principal Investigator — Virginia Spine Institute
Locations (1):
- Virginia Spine Institute, Reston, Virginia, United States